CLINICAL TRIAL: NCT03973827
Title: An Open Label, Parallel Single Centre Trial of Wharton's Jelly Derived Allogeneic Mesenchymal Stromal Cells Repeated Treatment to Preserve Endogenous Insulin Production in Adult Patients Diagnosed with Type 1 Diabetes
Brief Title: Wharton´s Jelly Derived Mesenchymal Stromal Cell Repeated Treatment of Adult Patients Diagnosed with Type I Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NextCell Pharma Ab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProTrans-Repeat; 2018-004158-11 (EudraCT Number)
Record Dates: First submitted 2019-05-16; First posted 2019-06-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type1diabetes
Keywords: type 1 diabetes; diabetes; MSC's; Mesenchymal; Stem Cells; Stromal; Wharton´s Jelly
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose (Experimental): 3 patients receiving low dose
  Interventions: Drug: ProTrans
- Medium dose (Experimental): 3 patients receiving medium dose
  Interventions: Drug: ProTrans
- High dose (Experimental): 3 patients receiving high dose
  Interventions: Drug: ProTrans
- Control (Other): 6 patients
  Interventions: Other: Control

INTERVENTIONS:
Drug: ProTrans — Single infusion of 25, 100 or 200 million cells per patient.
  Other Names: Allogeneic transplantation with WJMSCs
  Arms: High dose; Low dose; Medium dose
Other: Control — No intervention. Control subjects.
  Arms: Control

SUMMARY:
An open label, parallel single centre trial of Wharton's Jelly derived allogenic mesenchymal stromal cells repeated treatment to preserve endogenous insulin production in adult patients diagnosed with type 1 diabetes

DETAILED DESCRIPTION:
This is a phase (I)/II study, and the purpose of this study is to determine whether, in adult patients diagnosed for type 1 diabetes, a repeated allogeneic infusion of WJMSCs is safe and to study changes in beta-cell function, metabolic control and Diabetes Treatment Satisfaction. The study population will consist of 15 adult male patients, 18-41 years of age (inclusive at both ends) diagnosed (<3,5 years) with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. A new written informed consent for participation of the study is required to be given before undergoing any study-specific procedures.
2. Only patients that have previously been dosed by the IMP according to protocol Protrans-1 are eligible for a second dose of Protrans.
3. No identified IMP related on-going adverse event, neither history of any adverse event that is evaluated potentially to be related to the previous IMP dosing in Protrans I.
4. Clinical history compatible with type 1 diabetes diagnosed less than 3 years before enrolment. This also includes control patients not receiving IMP.
5. Only male patients between 18-41 years of age will be included.
6. Mentally stable and, in the opinion of the investigator, able to comply with the procedures of the study protocol.

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients with body mass index (BMI) > 30, or weight >100 kg
3. Patients with weight <50 kg
4. Patients with unstable cardiovascular status incl. NYHA class III/IV or symptoms of angina pectoris.
5. Patients with uncontrolled hypertension (≥160/105 mmHg).
6. Patients with active on-going infections.
7. Patients with latent or previous as well as on-going therapy against tuberculosis, or exposed to tuberculosis or has travelled in areas with high risk of tuberculosis or mycosis within the last 3 months.
8. Patients with serological evidence of infection with HIV, Treponema pallidum, hepatitis B antigen (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.
9. Patients with any immune suppressive treatment
10. Patients with known demyelinating disease or with symptoms or physical examination findings consistent with possible demyelinating disease.
11. Patients with known, or previous, malignancy.
12. Taking oral anti-diabetic therapies or any other concomitant medication which may interfere with glucose regulation other than insulin
13. Patients with GFR <80 ml/min/1.73 m2 body surface
14. Patients with proliferative retinopathy
15. Patient with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo treatment with MSC.
16. Known hypersensitivity against any excipients, i.e. dimethyl sulfoxide (DMSO).- This criterion is only applicable to patients which receive study drug.

Ages: 18 Years to 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this study is; safety parameters include adverse events and hypoglycemia, allergic reactions, ophthalmologic examination, ECG, vital signs, laboratory assessments. | 372 days
  To investigate the safety and tolerance after a repeated allogeneic infusion of Whartons Jelly Mesenchymal Stromal Cells (WJMSCs) intravenously in adult patients diagnosed with type 1 diabetes after one year following the repeated treatment.
Delta-change of C-peptide AreaUnder the Curve (AUC) (0-120 min) for Mixed Meal Tolerance Test (MMTT) at day 372 following WJMSC infusion when compared to test performed before start of treatment when compared to control patients. | 372 days
  To study changes in insulin requirements during one year following treatment .

SECONDARY OUTCOMES:
Number of patients insulin independent (ADA criteria) at day 372. | 372 days
  To study changes in insulin requirements during one year following treatment .
Number of patients with daily insulin needs <0.25U/kg at day 372. | 372 days
  To study changes in insulin requirements during one year following treatment .
Insulin requirement/kg BW at day 372. HbA1c at day 372. | 372 days
  To study changes in insulin requirements during one year following treatment .
HbA1c at day 372 | 372 days
  To study changes in HbA1c during one year following treatment.
Glucose variability (mean amplitude of glycaemic excursions and glycaemic lability index) duration derived from the continuous glucose monitoring system® at day 372 | 372 days
  To study changes in glucose levels during one year following treatment.
Delta change of levels of fasting C-peptide at day 372 when compared to test before start of treatment | 372 days
  To study changes in fasting C-peptide levels during one year following treatment.
Numbers of patients with peak C-peptide >0.20 nmol/l, in response to the MMTT, at day 372. | 372 days
  To study changes in C-peptide levels during one year following treatment.
To study changes during one year following treatment in: -Insulin doses -HbA1c -Glucose variability -Diabetes Treatment Satisfaction | 372 days
  To study changes in C-peptide levels during one year following treatment.
To study changes in insulin requirements during one year following treatment | 372 days
  2. Delta-change of C-peptide AreaUnder the Curve (AUC) (0-120 min) for Mixed Meal Tolerance Test (MMTT) at day 372 following WJMSC infusion when compared to test performed before start of treatment when compared to control patients.
  Description:

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, PhD, Principal Investigator — Uppsala University
Locations (1):
- Karolinska Trial Alliance, Fas 1 enheten, Karolinska Universitetssjukhuset Huddinge, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No